CLINICAL TRIAL: NCT01481623
Title: Identification and Genetic, Clinical and Metabolic Characterization of Monogenic Forms of Insulin-dependent Diabetes
Brief Title: Identification and Characterization of Monogenic Diabetes
Acronym: DIAGENE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P081230
Record Dates: First submitted 2011-10-27; First posted 2011-11-29 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes
Keywords: Diabetes; neonatal; consanguinity; monogenic; metabolism
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gene identification and phenotyping (Other): Identification of patients (probands), questionnaire and informed consent of patients and their families, biological sampling, DNA and RNA extraction, genetic study for gene identification, re-contact of family members and relatives (with consent) for metabolic study of mutation carriers, and complementary studies of homozygous patients in some cases
  Interventions: Other: Constitution of a biological bank; Other: Metabolic studies

INTERVENTIONS:
Other: Constitution of a biological bank — Blood samples for the constitution of a biobank (DNA, RNA, serum)
Other: Metabolic studies — oral glucose tolerance test (OGTT) intravenous glucose tolerance test (IVGTT) hyperglycemic clamp staged glucose perfusion arginine test measure of body composition (BIPHOTONIC absorptiometry, DEXA)

SUMMARY:
Type 1 Diabetes is a multifactorial disease, with a strong genetic contribution of HLA genes, and minor contributions of many additional genes. The investigators hypothesis is that in addition to multifactorial inheritance, there are subtypes of diabetes that are caused by defects in single genes (monogenic diabetes). The aim of this project is to identify these genes, based on detailed clinical and characterization of patients, and to describe the corresponding genetic diabetes entities with respect to the genetic and molecular defect, clinical features and biochemistry. Based on the investigators study design, most of these diabetes entities will be caused by mutations affecting the two copies of the corresponding gene. In addition, the investigators will study the relatives of the patients, and explore if carriers of these genetic defects (i.e. only one copy of the gene being defective) may have a predisposition to common forms of diabetes, mainly type 2 diabetes.

DETAILED DESCRIPTION:
In the first phase of the study the investigators will recruit patients and families, with a strong bias for "extreme" forms of diabetes (very early onset and/or syndromic diabetes) and familial context suggestive of monogenic inheritance (e.g. consanguinity, multiplicity of diabetic siblings) and perform genetic studies on these to identify the genes. After obtaining informed consent, the investigators will collect clinical information on diabetes and other associated diseases and features, family information on diabetes, and collect blood samples for DNA, RNA, serum and cell lines. The investigators will then perform genetic studies to identify the genes responsible for these monogenic forms of diabetes.

After identification of genes, the second phase of the study will be to test the consequence of carrier status for the identified mutations on metabolic traits related to glucose metabolism. For this, after obtaining informed consent, the investigators will extend the recruitment of the initial families (after gene identification) to recruit relatives who may be carriers of these mutations. The investigators will determine the carrier status of these subjects and perform a detailed clinical description as well as metabolic studies to evaluate their glucose metabolism.

This study will lead to the identification of new monogenic diabetes entities, and their corresponding genes, and may also result in the identification of new genes predisposing to common forms of diabetes. This project has implication for diagnosis of these monogenic forms of diabetes, and may result in some cases in improved care for the patients, including prevention and treatment.

ELIGIBILITY:
Inclusion Criteria:

* First phase: to have an "extreme" form of diabetes, based on clinical, phenotypic and familial criteria. Parents and siblings of the proband will be sampled.
* Second phase: (after gene identification): to be a relative of the proband, potential carrier of the mutation

Exclusion Criteria:

* Non consent to participate to the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Identification and genetic, clinical and metabolic characterization of monogenic diabetes forms | 36 months
  to identify genes responsible for monogenic insulin-dependant diabetes, and to define and characterize the corresponding genetic diabetes entities with respect to the genetic and molecular defect, clinical and phenotypic features and biochemistry

SECONDARY OUTCOMES:
Diagnosis of monogenic diabetes | 36 months
  to diagnose these monogenic diabetes entities and to evaluate the proportion of insulin-dependant diabetes which are explained by monogenic determinism, depending on several parameters, such as familial structure and clinical characteristics.
Clinical and biological characterization of total or partial deficiency of the genes responsible for monogenic diabetes | 36 months
  To characterize precisely the clinical and biological consequences of total or partial deficiency of the genes responsible for monogenic diabetes, and explore their possible role in glucidic metabolism. This way suggest them as candidate genes for common forms of diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Jean Guillausseau, MD, Study Director — CHU Lariboisière, AP-HP
Locations (1):
- Lariboisiere hospital, Paris, France